CLINICAL TRIAL: NCT03220425
Title: A Six Month, Multi-centre, Open-label, Parallel Efficacy and Safety Comparison of Insulin Detemir and NPH Insulin in Subjects With Type 1 Diabetes on a Basal-bolus Regimen.
Brief Title: Evaluation of the Efficacy and Safety of Insulin Detemir Compared With That of NPH Insulin in Subjects With Type 1 Diabetes.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NN304-1335
Record Dates: First submitted 2017-07-13; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Insulin detemir (Experimental)
  Interventions: Drug: Insulin detemir
- NPH insulin (Active Comparator)
  Interventions: Drug: NPH insulin

INTERVENTIONS:
Drug: Insulin detemir
  Arms: Insulin detemir
Drug: NPH insulin
  Arms: NPH insulin

SUMMARY:
The aim of this trial is to evaluate the efficacy and safety of insulin detemir using the 2400 nmol/mL formulation to optimise dosing in subjects with type 1 diabetes on a basal (once daily)-bolus regimen.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained before any trial-related activities
* Type 1 diabetes diagnosed and classified according to aetiology
* Duration of type 1 diabetes equal to or more than 12 months
* Glycosylated haemoglobin less than or equal to 12 percent based on analysis from central laboratory
* Able and willing to perform self-blood glucose monitoring

Exclusion Criteria:

* Proliferative retinopathy
* Total basal insulin dose of more than 100 IU per day
* Recurrent major hypoglycaemia - that would interfere with trial participation (as judged by the investigator)
* Known unawareness of hypoglycaemia
* Previous treatment with insulin detemir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2001-02-01 (Actual); Primary Completion 2001-11-12 (Actual); Study Completion 2001-11-12 (Actual)

PRIMARY OUTCOMES:
The change in the level of glycosylated haemoglobin(HbA1c) | From start of treatment visit 2 (week 0) until end of treatment visit 8 (week 26)

CONTACTS AND LOCATIONS:
Locations (88):
- Australia (8):
  - Novo Nordisk Investigational Site, Broadmeadow, New South Wales
  - Novo Nordisk Investigational Site, Ashford
  - Novo Nordisk Investigational Site, Box Hill
  - Novo Nordisk Investigational Site, Clayton
  - Novo Nordisk Investigational Site, Garran
  - Novo Nordisk Investigational Site, Ringwood
  - Novo Nordisk Investigational Site, Stones Corner
  - Novo Nordisk Investigational Site, Woodville
- Belgium (5):
  - Novo Nordisk Investigational Site, Bornem
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Ghent
  - Novo Nordisk Investigational Site, Leuven
  - Novo Nordisk Investigational Site, Luxembourg
- Denmark (8):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Copenhagen
  - Novo Nordisk Investigational Site, Fredericia
  - Novo Nordisk Investigational Site, Frederiksberg
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, Middelfart
  - Novo Nordisk Investigational Site, Odense
  - Novo Nordisk Investigational Site, Vejle
- Finland (5):
  - Novo Nordisk Investigational Site, Espoo
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Joensuu
  - Novo Nordisk Investigational Site, Kemi
  - Novo Nordisk Investigational Site, Vantaa
- France (12):
  - Novo Nordisk Investigational Site, Angers
  - Novo Nordisk Investigational Site, Avignon
  - Novo Nordisk Investigational Site, Bondy
  - Novo Nordisk Investigational Site, Corbeil-Essonnes
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Poitiers
  - Novo Nordisk Investigational Site, Rennes
- Novo Nordisk Investigational Site, Dublin, Ireland
- Netherlands (8):
  - Novo Nordisk Investigational Site, Amersfoort
  - Novo Nordisk Investigational Site, Apeldoorn
  - Novo Nordisk Investigational Site, Brunssum
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Haarlem
  - Novo Nordisk Investigational Site, Hengelo
  - Novo Nordisk Investigational Site, The Hague
  - Novo Nordisk Investigational Site, Utrecht
- Norway (8):
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Jessheim
  - Novo Nordisk Investigational Site, Kongsvinger
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Sarpsborg
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Stord
  - Novo Nordisk Investigational Site, Trondheim
- Sweden (10):
  - Novo Nordisk Investigational Site, Falun
  - Novo Nordisk Investigational Site, Helsingborg
  - Novo Nordisk Investigational Site, Karlstad
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Örebro
  - Novo Nordisk Investigational Site, Skövde
  - Novo Nordisk Investigational Site, Stockholm
  - Novo Nordisk Investigational Site, Umeå
  - Novo Nordisk Investigational Site, Uppsala
  - Novo Nordisk Investigational Site, Värnamo
- United Kingdom (23):
  - Novo Nordisk Investigational Site, Abergavenny
  - Novo Nordisk Investigational Site, Blackburn
  - Novo Nordisk Investigational Site, Bolton
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Cosham
  - Novo Nordisk Investigational Site, Derby
  - Novo Nordisk Investigational Site, Gillingham
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Kettering
  - Novo Nordisk Investigational Site, Livingstone
  - Novo Nordisk Investigational Site, Llantrisant
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Newcastle
  - Novo Nordisk Investigational Site, Northampton
  - Novo Nordisk Investigational Site, Norwich
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Sidcup
  - Novo Nordisk Investigational Site, Stevenage
  - Novo Nordisk Investigational Site, Taunton
  - Novo Nordisk Investigational Site, York

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk Disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Russell-Jones D, Simpson R, Hylleberg B, Draeger E, Bolinder J. Effects of QD insulin detemir or neutral protamine Hagedorn on blood glucose control in patients with type I diabetes mellitus using a basal-bolus regimen. Clin Ther. 2004 May;26(5):724-36. doi: 10.1016/s0149-2918(04)90072-0. PMID 15220016